CLINICAL TRIAL: NCT06961760
Title: A Single-arm, Open-label, Expanded Access Program to Provide 100 mg CT1812 (Zervimesine) and to Collect Long-term Safety and Efficacy Data in Participants With Mild-to-moderate Dementia With Lewy Bodies (DLB).
Brief Title: Expanded Access Program for CT1812 (Zervimesine)
Status: No longer available | Type: Expanded Access
Sponsor: Cognition Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: COG1202
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Dementia With Lewy Bodies
Keywords: Dementia
MeSH Terms: conditions — Lewy Body Disease; Dementia

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: zervimesine — Zervimesine (CT1812) was shown to be safe and well tolerated in a study of healthy volunteers and in Phases 1 and 2 studies of participants with mild to moderate AD and DLB. This is an open label expanded access program designed to provide access to CT1812 and to evaluate the long-term safety of CT1812 administered once daily for 12 months in adults aged 50 to 86 who have been diagnosed with mild to moderate DLB (the targeted clinical indication for CT1812). Participants will receive 100 mg of CT1812 once daily for 360 days.
  Other Names: CT1812

SUMMARY:
This is a multi-center, open label, expanded access program (EAP) that will provide 100 mg CT1812 for up to one year to participants with mild-to-moderate DLB.

DETAILED DESCRIPTION:
Participants will be screened for eligibility by physical, laboratory, psychometric and neurologic examinations. After having met all inclusion criteria, and none of the exclusion criteria, participants will be enrolled. The first dose will be taken in the clinic. Participants and their caregivers/study partner will have a study visit clinic for repeat psychometric/neurologic testing, safety procedures and lab sample collection. Each participant and caregiver/study partner will participate in a screening period of up to 7 days, followed by an open label treatment period of 360 (± 4 days) days and a follow up visit at day 390 (± 2 days) for a maximum of 397 days of study participation including screening.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must meet either one of the following criteria:

   1. Randomized participant in protocol COG1201 and completed the study or
   2. Referred by their treating physician to a participating COG1202 study site with a confirmed diagnosis of DLB, provide evidence of a historical MRI (within last 3 months) or CT-Scan (within last 3 months), a baseline Mini Mental Status Examination score (MMSE) of 18 - 27 inclusive and be approved by Sponsor
2. Participants must have caregiver(s) / study partner who in the opinion of the site principal investigator, has contact with the study participant for a sufficient number of hours per week to provide informative responses on the protocol assessments, oversee the administration of study drug, and willing and able to participate in study visits and some study assessments. The caregiver/ study partner must also provide informed consent to participate in the study.
3. Men or women 50- 86 years of age (inclusive).
4. Must have had no clinically relevant findings, other than change for progression of DLB, on historical MRI or CT scan.
5. In the opinion of the investigator, must be able to complete all protocol evaluations.

Exclusion Criteria:

1. If enrolled in the previous CT1812 clinical trial for DLB (COG1201), did not complete the clinical trial, or had an adverse event that could cause an undue risk, or progressed to severe DLB and cannot complete study assessments.
2. Any neurological condition that may be contributing to cognitive impairment and beyond those caused by the participant's DLB.
3. History of cancer within 3 years of screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months based on imaging or Prostate-Specific Antigen (PSA) levels.
4. Clinically significant, advanced or unstable disease that may interfere with outcome evaluations.
5. Any condition, which in the opinion of the investigator or the sponsor makes the participant unsuitable for inclusion.
6. No access to a Primary Care Physician, inability or unwillingness to have lab sample collection completed per protocol.

Ages: 50 Years to 86 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, PHD, Study Director — Cognition Therapeutics Inc.
Locations (8):
- United States (8):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Stanford Neuroscience Heath Center, Palo Alto, California
  - University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado
  - University of Miami - Department of Neurology, Boca Raton, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Ohio State University Wexner Medical Center (OSUWMC), Columbus, Ohio
  - Summit Headlands LLC, Portland, Oregon